CLINICAL TRIAL: NCT06676969
Title: Evaluation of High and Low Flow Sevoflurane Anesthesia in Pediatric Patients Undergoing Laparoscopic Surgeries in Terms of Recovery, Hemodynamics, and Cost
Brief Title: High vs. Low Flow Sevoflurane Anesthesia in Pediatric Laparoscopic Surgery: Recovery, Hemodynamics, and Cost Comparison
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sibel Barış, Professor, Ondokuz Mayıs University
Other Study IDs: High/Low flow Anestesia
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Low-flow Anesthesia
Keywords: Laparoscopic surger; Low-flow anesthesia; Pediatric Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low flow: Low flow Anestesia
- High Flow: High Flow Anestesia

SUMMARY:
The primary objective of our study is to compare the effects of different flow rates of the routinely used inhalation agent, sevoflurane, on postoperative recovery times in pediatric patients undergoing elective laparoscopic surgeries. Our secondary objectives are to evaluate the impact of different flow rates on hemodynamic parameters, ventilation parameters, and costs.

DETAILED DESCRIPTION:
Low-flow anesthesia is a technique in which at least 50% of the exhaled gas is returned to the system through rebreathing. When using modern rebreathing systems, low-flow anesthesia can be defined if the fresh gas flow rate is reduced below 2 L/min. This anesthesia method involves using an anesthesia system with rebreathing capabilities, where carbon dioxide is removed from the gas mixture exhaled by the patient, and then at least 50% of the fresh oxygen flow, along with volatile anesthetics sufficient to meet the body's metabolic requirements, is returned to the patient.

The application of low-flow anesthesia reduces the consumption of anesthetic gases, decreases the cost of anesthesia, minimizes contamination of the working environment and atmosphere with anesthetic gases, preserves the respiratory physiology of the patient, and minimizes heat and humidity loss by heating and humidifying the gases delivered to the patient, thereby better maintaining the physiology of the trachea and bronchial environments. The heating of gases is also beneficial for maintaining body temperature and preventing postoperative hypothermia. Additionally, due to the requirement for close monitoring, anesthesia safety is increased .

In pediatric patients, due to their different anatomical and physiological characteristics compared to adults, the application of low fresh gas flow anesthesia can be more challenging. This is especially the case when using uncuffed endotracheal tubes, where leaks may occur in the respiratory system, and the breathing circuits used may increase dead space. However, studies have shown that with appropriate techniques and adequate monitoring, these potential problems can be prevented, and low-flow anesthesia can be safely applied in children with close monitoring.

In our study, the investigators aim to compare the effects of different flow rates on postoperative recovery, hemodynamic factors, and costs in children, and to demonstrate that low-flow anesthesia can be applied as safely as high-flow anesthesia in pediatric patients. The investigators believe our study will contribute significantly to the literature on this topic.

ELIGIBILITY:
Inclusion criteria:

Patients with an American Society of Anesthesiologists (ASA) classification of I-II.

Elective laparoscopic surgeries expected to last longer than 30 minutes but shorter than 180 minutes

Exclusion Criteria:

Patients who are not candidates for laparoscopic surgery. Patients unsuitable for low-flow anesthesia due to inadequate monitoring conditions.

Patients whose relatives are unable to provide informed consent. Patients with an American Society of Anesthesiologists (ASA) classification higher than II.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients undergoing laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Recovery times with Aldrete recovery score | 15/09/24-30/11/24

SECONDARY OUTCOMES:
Incidence of intraoperative hypothermia by esophageal temperature measurements | 15/09/24-30/11/24

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - 19 Mayis Üniversitesi Tip Fakültesi, Samsun
  - 19 Mayıs Üniversitesi Tıp Fakültesi, Samsun

REFERENCES:
- [Background] Isik Y, Goksu S, Kocoglu H, Oner U. Low flow desflurane and sevoflurane anaesthesia in children. Eur J Anaesthesiol. 2006 Jan;23(1):60-4. doi: 10.1017/S026502150500178X. PMID 16390568
- [Background] Park SY, Chung CJ, Jang JH, Bae JY, Choi SR. The safety and efficacy of minimal-flow desflurane anesthesia during prolonged laparoscopic surgery. Korean J Anesthesiol. 2012 Dec;63(6):498-503. doi: 10.4097/kjae.2012.63.6.498. Epub 2012 Dec 14. PMID 23277809
- [Background] Glenski TA, Levine L. The implementation of low-flow anesthesia at a tertiary pediatric center: A quality improvement initiative. Paediatr Anaesth. 2020 Oct;30(10):1139-1145. doi: 10.1111/pan.13994. Epub 2020 Aug 29. PMID 32786105
- [Background] Meakin GH. Low-flow anaesthesia in infants and children. Br J Anaesth. 1999 Jul;83(1):50-7. doi: 10.1093/bja/83.1.50. No abstract available. PMID 10616333
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/